CLINICAL TRIAL: NCT00219791
Title: Study of Recombinant Carboxypeptidase G2 (CPG2) for the Management of Patients With Delayed Methotrexate (MTX) Clearance or Intrathecal MTX Overdosage
Brief Title: Study of Glucarpidase (CPG2) for the Management of Patients With Delayed Methotrexate Clearance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BTG International Inc. (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR001-CLN-rpt002; ek.179-6
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Neoplasms
Keywords: methotrexate; delayed elimination; renal insufficiency; CPG2; Voraxaze
MeSH Terms: conditions — Neoplasms; Renal Insufficiency | interventions — glucarpidase

INTERVENTIONS:
Drug: glucarpidase (50 Units/kg)

SUMMARY:
To evaluate the safety and efficacy of glucarpidase in patients with impaired methotrexate (MTX) clearance owing to MTX-induced renal failure following high-dose MTX therapy, or with intrathecal MTX overdose.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by patient or legally valid representative
* Patients receiving high-dose MTX (>1 g/m2 body surface area (BSA) given as an infusion over 24 hours) for the treatment of ALL, NHL or a solid tumour (e.g. osteosarcoma)
* Age ≥ 18 years
* Serum MTX >5 µmol/L 42 hours or later after the start of MTX infusion, or serum MTX >1 μmol/L 42 hours or later after the start of MTX infusion together with renal insufficiency, or serum MTX >0.4 µmol/L 48 hours or later after the start of MTX infusion together with renal insufficiency. Renal insufficiency was defined as serum creatinine >1.5 × the upper limit of normal (ULN) and/or oliguria (urine output < 500 mL/24 hours despite adequate hydration, diuretics and alkalinisation).

Exclusion Criteria:

* Pregnant or lactating females
* Unwillingness of patient or relative/legal representative to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Study Completion 2003-06

PRIMARY OUTCOMES:
Reduction in serum MTX concentration

SECONDARY OUTCOMES:
serum blood-urea-nitrogen
serum creatinine
creatinine clearance
haematology (complete blood count and differential)
biochemistry (electrolytes, SGOT, SGPT, alkaline phosphatase, bilirubin, total protein)
urinalysis (dip-stick)
MTX-related toxicity
Adverse events
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Thiel Eckhard, Prof. Dr.med., Principal Investigator — Charite - Universitätsmedizin Berlin
Locations (1):
- Charite - Universitätsmedizin Berlin, Berlin, Germany